CLINICAL TRIAL: NCT06748404
Title: A Phase 2 Randomized Study of TriCalm Hydrogel® in the Treatment of Immunotherapy-Related Pruritus
Brief Title: TriCalm Hydrogel® in the Treatment of Immunotherapy-Related Pruritus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Karen Yun, Assistant Clinical Professor, Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 809201
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Immunotherapy-related Pruritus
Keywords: Immunotherapy; Pruritus
MeSH Terms: conditions — Pruritus | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: This is a phase 2, randomized, open-label, single-center clinical trial that will assess the efficacy of TriCalm Hydrogel® in treating pruritus related to immune checkpoint inhibitors (ICIs). Patients will be randomized 1:1 to receive 2 cycles of TriCalm Hydrogel® versus one cycle of topical corticosteroid followed by one cycle of TriCalm Hydrogel®. A randomized comparison of the change in mean Numeric Rating Scale (NRS) scores between each treatment arm will be performed. Patients will be stratified by 3-week and 4-week ICI cycles. Efficacy and safety outcomes will be assessed over a period of 2 cycles of ICI therapy ranging 6-8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A (Experimental): TriCalm Hydrogel® during cycles 1 and 2
  Interventions: Drug: Tricalm Hydrogel
- ARM B (Active Comparator): Triamcinolone cream during cycle 1 followed by Tricalm Hydrogel® during cycle 2
  Interventions: Drug: Tricalm Hydrogel; Drug: Triamcinolone acetonide 0.1% cream

INTERVENTIONS:
Drug: Tricalm Hydrogel — TriCalm Hydrogel® is a topical gel that allows rapid administration to areas of the skin. TriCalm Hydrogel® is available over-the-counter and contains the active ingredient, aluminum acetate 0.2%, and inactive ingredient, strontium chloride hexahydrate.
  Other Names: TriCalm Steroid Free Soothing Itch Relief Hydrogel
Drug: Triamcinolone acetonide 0.1% cream — Triamcinolone acetonide 0.1% cream is a topical steroid cream that will be applied directly to the skin.
  Other Names: Triamcinolone Acetonide
  Arms: ARM B

SUMMARY:
This is a phase 2, randomized, open-label, single-center study that will assess the efficacy of TriCalm Hydrogel®, a topical gel containing strontium, for treating pruritus related to immune checkpoint inhibitors (ICIs).

DETAILED DESCRIPTION:
Pruritus is a common immune-related adverse event of immune checkpoint inhibitors (ICI).

This is a phase 2, randomized, open-label, single-center study that will assess the efficacy of TriCalm Hydrogel®, a topical gel containing strontium, for treating pruritus related to ICIs. Topical strontium salts have been found to reduce the duration and severity of histaminergic and nonhistaminergic pruritus. The investigators hypothesize that TriCalm Hydrogel® will be effective in reducing the severity of immunotherapy-related pruritus and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Patients receiving ICIs for hematologic or oncologic malignancies at the Moores Cancer Center Infusion Center at UC San Diego. ICIs include CTLA-4 inhibitors (ipilimumab), PD-1 inhibitors (cemiplimab, nivolumab, pembrolizumab) and PD-L1 inhibitors (atezolizumab, avelumab, durvalumab).
3. Patients who develop grade 1-3 pruritus at any time after receiving at least one dose of ICI.
4. Preexisting use of oral antihistamines and/or GABA analogs more than 7 days prior to study entry are allowed.

Exclusion Criteria:

1. Diagnosis of primary skin disorders with pruritus symptoms (e.g., atopic dermatitis, psoriasis).
2. Initiation of any new oral or topical antipruritic medications and/or systemic corticosteroids within 7 days prior to study entry.
3. Presence of open wounds on the skin.
4. Presence of pruritus on the face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of TriCalm Hydrogel® in reducing the severity of immunotherapy-related pruritus. | 6-8 weeks
  Efficacy of TriCalm Hydrogel® in reducing the severity of pruritus as defined as change in mean pruritus Numeric Rating Scale (NRS) scores.
  A randomized comparison of the change in mean pruritus NRS scores after cycle 1 (Arm A, one cycle of TriCalm Hydrogel®; Arm B, one cycle of topical corticosteroid) will be tested between treatment arms.
  NRS is a single item questionnaire assessing the patient-reported severity of itch at its greatest intensity over the past 24 hours on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'the worst itch'. NRS scores will be assessed weekly in this study.

SECONDARY OUTCOMES:
To evaluate the efficacy of TriCalm Hydrogel® in improving the quality of life in patients with immunotherapy-related pruritus. | 6-8 weeks
  Change in mean Dermatology Life Quality Index (DLQI) scores after 1 and 2 cycles of TriCalm Hydrogel® for all patients in both treatment arms will be assessed by 95% confidence intervals.
  Randomized comparison of the change in mean pruritus DLQI scores, after cycle 2, between treatment arms will be assessed by 95% confidence intervals.
  DLQI is a 10-item questionnaire assessing the impact of pruritus on quality of life in the last 7 days. Responses are scored on a 4-point scale ranging from 0 (not at all or not relevant) to 3 (very much) for a total maximum of 30 points and a minimum of 0 points. Higher total scores correspond to greater impairment in quality of life. DLQI scores will be assessed weekly in this study.
To evaluate the safety of TriCalm Hydrogel® in patients with immunotherapy-related pruritus. | 6-8 weeks
  Adverse events (AEs) related to TriCalm Hydrogel®. AEs will be graded according to CTCAE version 5.0. Incidence, description, timing, severity, and relatedness of AEs will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Yun, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No